CLINICAL TRIAL: NCT00966680
Title: Speed of General Versus Spinal Anesthesia for Emergency Cesarean Delivery: A Simulation Based Study
Brief Title: How Fast Are we? Speed of General Versus Spinal Anesthesia for Emergency Cesarean Delivery: A Simulation Based Study
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H09-01465
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Anesthesia
Keywords: general anesthesia; spinal anesthesia; emergency cesarean delivery
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — 16 anesthesiologists will be recruited for the simulation part. 100 women having elective cesarean delivery will be timed in the clinical part.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Observational study comparing the speed of general versus spinal anesthesia during emergency cesarean
  Interventions: Other: Anesthesia

INTERVENTIONS:
Other: Anesthesia — How long anesthesiologists take to administer general and spinal anesthesia.

SUMMARY:
The researchers wish to undertake a simulation based study to compare the speed of general versus spinal anesthesia for emergency cesarean delivery. Minutes may matter for the baby in an emergency. It is unknown which technique is quicker. Their hypothesis is that surgical anesthesia can be achieved as quickly with spinal as with general anesthesia.

DETAILED DESCRIPTION:
Rapid delivery of the fetus by emergency cesarean delivery is usually necessary when there is risk to mother or fetus (1). Some maternal indications for emergency cesarean delivery include uncontrolled bleeding, high spinal block and cardiac arrest. For the fetus, minutes may count when there are abnormal fetal heart rate patterns such as accompanying uterine rupture or umbilical cord prolapse. Under these emergency circumstances published recommendations include that delivery should occur within 30 minutes from decision time (2). Thus, the time taken to achieve surgical anesthesia is important and should be kept as short as possible to minimize risk to the fetus (3).

In the absence of a pre-existing labor epidural that can be rapidly extended for anesthesia, general (GA) or spinal (SA) anesthesia are usually administered to facilitate delivery in the urgent/emergent situation. Each technique has risks and benefits, but the choice of anesthesia will ultimately depend upon the circumstances. For example, severe maternal bleeding would favor GA because it is perceived to be quicker (although there are no studies to confirm this) and uncontrolled hemorrhage can produce hemodynamic instability which can be exacerbated by SA. On the other hand, known reactions to anesthetic agents (such as malignant hyperthermia) would make SA more favorable.

There is a perception amongst anesthesiologists that GA in pregnant women is associated with increased morbidity and mortality. This is partly due to the increased use of regional anesthesia since the 1960s and the uncommon occurrence of general anesthesia has lead to increased incidence of complications worldwide (4, 5). The reasons for this relate to the physiological changes of pregnancy which can make endotracheal intubation more difficult, increase the risk of pulmonary aspiration of stomach contents and awareness of intraoperative events (6, 7). These potential risks mean that fewer general anesthetics for cesarean delivery are being done while numbers of central neuraxial blocks (spinal, epidural) have increased. This means that anesthesiologists are less experienced in general anesthesia for obstetrics (8, 9). As well, at delivery the infant is more likely to be initially depressed and require active resuscitation than those delivered by SA (10). The depression is due not only to the GA but also to the reason for rapid delivery, for example cord prolapse causing fetal distress.

Apart from avoiding the risks of GA, SA has the added advantage that the parturient is awake when the infant is born and can be accompanied by their partner in the OR. As morphine is given with the spinal medication the women will generally have less pain post-operatively as well as being clear minded. However, occasionally SA can fail necessitating a GA.

It is unknown which technique is quicker. Some anesthesiologists believe that SA can be administered as quickly as GA and will often persist in administering SA for fear of the risks of general anesthesia. However, after induction of general anesthesia and endotracheal intubation, surgery can start immediately while with SA surgical anesthesia takes some time to develop after the anesthetic drugs are injected. There are no studies examining when surgery can actually start following SA and GA. Direct comparison of the two techniques under emergency situations based on a randomized control trial is impossible due to problems obtaining consent in that emergency situation where minutes count. Marx et al found that spinal anesthesia can be induced as quickly as GA, but the spinal needle used was bigger and the drug used (amethocaine) is not commonly used in modern practice (11).

Simulation of emergency scenarios allows anesthesiologists to practice safe emergency anesthesia (12). In a pilot simulation study insertion of SA was found to be as quick as GA, but the time to achieve surgical anesthesia was longer (13). Thus, the overall time between inducing anesthesia and the time when surgery could actually start was longer with SA.

We wish to undertake a simulation based study to compare the speed of GA versus SA for emergency cesarean delivery. We also wish to observe the techniques anesthesiologists use to expedite readiness to surgical anesthesia. At the conclusion of this study, we hope to help the anesthesiologist decide upon the optimum technique of anesthesia for emergency cesarean delivery and so affect fetal and maternal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Consenting anesthesiologists,
* R5 residents and anesthesia fellows practicing at BC Women's Hospital

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consenting anesthesiologists, R5 residents and anesthesia fellows practicing at BC Women's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gunka, Dr., Principal Investigator — University of British Columbia; Arry Kathirgamanathan, Dr., Study Director — University of British Columbia; Roanne Preston, Dr., Study Director — University of British Columbia; Jessica Tyler, Ms., Study Director — University of British Columbia
Locations (1):
- BC Women's Hospital & Health Care, Vancouver, British Columbia, Canada